CLINICAL TRIAL: NCT02542618
Title: The Efficacy of Inquiry Based Stress Reduction (IBSR) for Depression, a Randomized Clinical Trial
Brief Title: The Efficacy of Inquiry Based Stress Reduction (IBSR) for Depression, a Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: FortaGroep (Unknown)
Responsible Party: Principal Investigator, Ingmar Franken, Professor of Clinical Psychology, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL51699.078.15
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Depression
Keywords: Depression; Treatment; IBSR; CBT
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inquiry Based stress Reduction (IBSR) (Experimental): IBSR intervention is the clinical implementation of a mindful-process, named "The Work" developed by Byron Katie. It teaches the individual to identify and question the thoughts that causes stress and suffering through four questions and turnarounds.
  Interventions: Behavioral: Inquiry Based Stress Reduction (IBSR)
- Cognitive Behavioral Therapy (CBT) (Active Comparator): CBT is a psychological treatment method, focusing on a structured way to identify and modify unhelpful thinking patterns, underlying assumptions and idiosyncratic cognitive schemes about the self, the world (including other people) and the future.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Inquiry Based Stress Reduction (IBSR)
  Other Names: The Work
  Arms: Inquiry Based stress Reduction (IBSR)
Behavioral: Cognitive Behavioral Therapy (CBT)
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
Background: Major depression is a common mental disorder with serious consequences. The societal costs of depression are high. Despite the existence of empirically-supported psychological therapies, many patients do not benefit from these treatments and relapse and recurrence percentages are high. Improvement of existing treatments or development of new and better treatments is badly needed. Inquiry Based Stress Reduction (IBSR) is a promising verbal therapy focusing on the inquiry of thoughts and could be a next step in improving psychotherapy for depression.

Objective: The objective of the current study is to assess the effectiveness of IBSR. Research to date has shown that IBSR is effective in reducing symptoms of anxiety and depression. The investigators want to know if IBSR is more effective in reducing symptoms of depression than the best psychotherapeutic treatment for depression at this moment, cognitive behavioural therapy (CBT). The investigators' secondary objective is to know more about the underlying mechanisms of change of these therapies.

Study design: A randomized controlled intervention study.

Study population: 88 patients with a mild to moderate depression as their principal diagnosis.

Intervention: IBSR or CBT

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older,
* Not making use of other treatment for depression at the time,
* No history of psychotherapy in the last year,
* No medication for depression or unchanged dosage of medication during the last two months ,
* All participants must be willing to refrain from engaging in additional psychological treatments or making changes to their medication status during the course of the trial. (changes in medication dosage will result in dropout),
* All participants must have at least a low average level of intelligence (IQ above 80). During regular intakes a clinical judgment is made. This is in accordance with the standard protocols used within the FortaGroep.
* All participants are required to have sufficient knowledge of the Dutch language.

Exclusion Criteria:

* Active suicidal intent (which is asked during the interviews and further operationalized with help of the ninth item in the BDI-II at pre-treatment: If patients marked the statement ''I would kill myself if I could'', they are classified as being at risk of suicide)
* If the DSM-IV criteria for severe major depressive disorder, psychotic disorder, or bipolar disorder are met
* A mental impairment or neurocognitive disorders such as Alzheimer
* Substance abuse requiring specialist treatment
* No time for homework.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-II) to measure change from baseline self-reported symptoms of depression at the endpoint of the therapy (after completing 16 sessions) and follow-ups. | At pre (baseline) and session 16 (post) and follow-up (after 1 and 2 years) measurements.
  The BDI-II is a self-report questionnaire which measures the severity of depression in 21 statements, with four levels of increasing severity each. The investigators use the BDI-II to measure self-reported symptoms of depression.

SECONDARY OUTCOMES:
Symptom Questionnaire (SQ-48) to measure change in self-reported general psychological distress from baseline at session 8, session 16 (end of therapy) and follow-ups | At pre (baseline), session 8 and 16 (post) and follow-up (after 1 and 2 years) measurements.
  The SQ-48 is a self-report questionnaire which measures general psychological distress, vitality/optimism and work functioning. The subscales of this questionnaire include: Depression, Anxiety, Somatization, Agoraphobia, Aggression, Cognitive problems, Social Phobia, Work functioning and Vitality. The investigators use the SQ-48 to measure general psychological distress.
Short Form Health Survey (SF-36) to measure change from baseline self-reported quality of life at the endpoint of the therapy (after completing 16 sessions) and follow-ups | At pre (baseline), session 16 (post) and follow-up (after 1 and 2 years) measurements.
  The SF-36 is a self-report questionnaire which measures quality of life. It consists of 36 items on well-being and functional, mental and physical health. The investigators use the SF-36 to measure quality of life.
The Structured Clinical Interview for Diagnostic and Statistical Manual-IV (DSM-IV) Axis I Disorders (SCID-I) Dutch version to screen for Diagnostic and Statistical Manual of Mental Disorder (DSM-IV) diagnoses | At pre (baseline), session 16 (post) and follow-up (after 1 and 2 years) measurements.
  This structured interview is used to determine DSM-IV Axis I disorders. The investigators use the SCID-I to check in- and exclusion criteria, and to determine change in diagnosis after therapy.
Acceptance and Action Questionnaire-II (AAQ-II) to measure change in self-reported level of general psychological acceptance from baseline at every fourth therapy session and follow-ups | At pre (baseline), session 4,8, 12 and 16 (post) and follow-up (after 1 and 2 years) measurements.
  The AAQ-II is a self-report questionnaire which measures the psychological acceptance component of psychological flexibility. The investigators use the AAQ-II to measure the level of general psychological acceptance.
Dysfunctional Attitude Scale, 17-item Dutch version (DAS-A-17) to measure change in self-reported level of dysfunctional thinking from baseline at every fourth therapy session and follow-ups | At pre (baseline), session 4,8, 12 and 16 (post) and follow-up (after 1 and 2 years) measurements.
  The DAS-A-17 is a self-report scale designed to measures the respondent's use of typical depressive assumptions. The investigators use the DAS-A-17 to measure the level of dysfunctional thinking.
Behavioral activation for depression scale (BADS) to measure change in self-reported level of activation from baseline at every fourth therapy session and follow-ups | At pre (baseline), session 4,8, 12 and 16 (post) and follow-up (after 1 and 2 years) measurements.
  The short version of the BADS is a self-report questionnaire which measures the amount of activation in the past week. The investigators use the BADS to measure the level of activation.
State-Trait Anxiety Inventory, version: Y (STAI-form Y) to measure the level of anxiety at baseline | At pre (baseline)
  The STAI assesses current and trait anxiety symptoms. The investigators use the STAI to measure anxiety at baseline.
Beck Depression Inventory (BDI-II) to measure change from baseline self-reported symptoms of depression at every fourth therapy session | At pre (baseline), session 4,8, 12 and 16 (post).

CONTACTS AND LOCATIONS:
Locations (1):
- FortaGroep, Rotterdam, South Holland, Netherlands